CLINICAL TRIAL: NCT04352140
Title: Electromyographic and Acceleromyographic Monitoring in Restricted Arm Movement Surgical Setting. A Prospective, Randomized Trial.
Brief Title: Electromyographic and Acceleromyographic Monitoring in Restricted Arm Movement Surgical Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, J. Ross Renew, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-000629
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Results first posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-01

CONDITIONS: Residual Neuromuscular Blockade
Keywords: Neuromuscular Blockade; Tetragraph; AMG; EMG
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Dominant hand (Experimental): Subject scheduled to undergo an elective surgical procedure will have TetraGraph device lead placement on the dominant hand, ToFscan placed on non-dominant hand
  Interventions: Device: Tetragraph; Device: ToFscan
- Non-dominant hand (Experimental): Subject scheduled to undergo an elective surgical procedure will have TetraGraph device lead placement on the non-dominant hand, ToFscan placed on dominant hand
  Interventions: Device: Tetragraph; Device: ToFscan

INTERVENTIONS:
Device: Tetragraph — FDA approved neuromuscular transmission monitor capable of measuring the depth of neuromuscular block in anesthetized patients who received neuromuscular blocking agents. TetraGraph uses EMG to measure the muscle action potentials that are generated in response to electrical neurostimulation via skin electrodes.
Device: ToFscan — ToFscan is a nerve stimulator module used for the measurement of neuromuscular transmission via accelerometry. ToFscan was developed by Drager Technologies, Canada, and it uses a three-dimensional piezoelectric sensor that attaches to the thumb via a hand adapter to measure acceleration in multiple planes (Murphy et al, 2018). Following simultaneous ulnar nerve stimulation on each arm, the response of the adductor pollicis will be measured

SUMMARY:
Researchers are comparing the ease of use and repeatability of the force vs electrical activity produced by a muscle after it has undergone nerve stimulation during a surgical procedure in which the patients' arm movement is restricted (placed under surgical drapes) in laparoscopic or robotic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years old
* Patients willing to participate and provide an informed consent
* Patients undergoing an elective laparoscopic or robotic surgical procedure that requires use of NMBA agents administered intraoperatively.

Exclusion Criteria:

* Patients with disorders, such as stroke, carpal tunnel syndrome, broken wrist with nerve damage, Dupuytren contracture, or any similar wrist injury.
* Patients with systemic neuromuscular diseases such as myasthenia gravis
* Patients with significant organ dysfunction that can significantly affect pharmacokinetics of neuromuscular blocking and reversal agents, i.e., severe renal impairment or end-stage liver disease.
* Patients having surgery that would involve prepping the arm or leg into the sterile field

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J.Ross Renew, MD, Principal Investigator — Mayo Clinic
Locations (3):
- Mayo Clinic in Florida, Jacksonville, Florida, United States
- Université de Lorraine, CHU de Brabois, Vandœuvre-lès-Nancy, France
- University of Debrecen, Debrecen, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Dominant Hand: Subject who received an elective surgical procedure had TetraGraph device lead placement on the dominant hand, ToFscan placed on non-dominant hand
  Tetragraph: FDA approved neuromuscular transmission monitor capable of measuring the depth of neuromuscular block in anesthetized patients who received neuromuscular blocking agents. TetraGraph uses EMG to measure the muscle action potentials that are generated in response to electrical neurostimulation via skin electrodes.
  ToFscan: ToFscan is a nerve stimulator module used for the measurement of neuromuscular transmission via accelerometry. ToFscan was developed by Drager Technologies, Canada, and it uses a three-dimensional piezoelectric sensor that attaches to the thumb via a hand adapter to measure acceleration in multiple planes (Murphy et al, 2018). Following simultaneous ulnar nerve stimulation on each arm, the response of the adductor pollicis will be measured
- Non-dominant Hand: Subject who received an elective surgical procedure had TetraGraph device lead placement on the non-dominant hand, ToFscan placed on dominant hand
  Tetragraph: FDA approved neuromuscular transmission monitor capable of measuring the depth of neuromuscular block in anesthetized patients who received neuromuscular blocking agents. TetraGraph uses EMG to measure the muscle action potentials that are generated in response to electrical neurostimulation via skin electrodes.
  ToFscan: ToFscan is a nerve stimulator module used for the measurement of neuromuscular transmission via accelerometry. ToFscan was developed by Drager Technologies, Canada, and it uses a three-dimensional piezoelectric sensor that attaches to the thumb via a hand adapter to measure acceleration in multiple planes (Murphy et al, 2018). Following simultaneous ulnar nerve stimulation on each arm, the response of the adductor pollicis will be measured
Period: Overall Study
Arm/Group | Dominant Hand | Non-dominant Hand
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dominant Hand | Non-dominant Hand | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (12.49) | 60.6 (14.04) | 60.37 (13.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 17 | 18 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 28 | 29 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 15 | 15 | 30
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Values Between Tetragraph and ToFscan
Description: The number of subject's who's residual neuromuscular blockage units are the same on both the TetraGraph and the ToFscan
Time Frame: Up to 1 hour postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Dominant Hand | Non-dominant Hand
Number analyzed (Participants) | 30 | 30
Participants | 0 | 2

2. Secondary Outcome: Incidence of Residual Neuromuscular Blockade
Description: Number of patients with train of four ratio < 0.9 after administration of reversal agent.
Time Frame: Up to 1 hour postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Dominant Hand | Non-dominant Hand
Number analyzed (Participants) | 30 | 30
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study for all subjects, approximately 1 hour
Arm/Group | Dominant Hand | Non-dominant Hand
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT04352140/Prot_SAP_000.pdf